CLINICAL TRIAL: NCT05210920
Title: RBG: Regular, Bare, Gel: Does Type of Nail Polish Affect Bacterial Counts After Surgical Scrubbing?
Acronym: RBG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-0027
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Bacterial Infections; Surgical Site Infection; Contaminated Medical or Biological Substances
MeSH Terms: conditions — Bacterial Infections; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: All participants will have all three nail types assessed: regular polish, gel polish and bare nail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular Nail Polish (Experimental): Participants will have regular nail polish applied to one fingernail of their dominant hand
  Interventions: Other: Nail polish application
- Gel Nail Polish (Experimental): Participants will have gel nail polish applied to one fingernail of their dominant hand
  Interventions: Other: Nail polish application
- Bare Nail (No Intervention): Participants will have one fingernail of their dominant hand left bare for comparison

INTERVENTIONS:
Other: Nail polish application — After application of nail polish as described, participants will have bacterial swabs collected from the under the fingernail and from the nail bed of the three assigned fingers on their dominant hand, both before and after scrubbing with a chlorhexidine surgical scrubbing brush.
  Arms: Gel Nail Polish; Regular Nail Polish

SUMMARY:
Purpose: The purpose of this study is to evaluate if type of nail polish (gel polish or regular polish) has an effect on the number of bacterial colonies on finger nails after surgical scrubbing.

Participants: The potential participants are healthcare providers with patient interaction. Exclusion criteria include evidence of active dermatitis or other skin abnormalities, or allergy to chlorhexidine.

Intervention: Participants will have gel nail polish applied to one finger of their dominant hand, and regular polish applied to another finger of their dominant hand. Bacterial swabs will be collected from these two fingers, as well as the from the adjacent finger with no nail polish. Specimen collection will occur both before and after scrubbing with surgical soap. Bacterial counts will be compared between the three groups to determine the association between the presence of nail polish and nail polish type on bacterial counts after surgical scrubbing. Specimen collection will not take place during scrubbing for actual patient care.

DETAILED DESCRIPTION:
Potential participants will be identified by word of mouth, flyers and institutional networking. Once a participant agrees to enroll, they will have each type of nail polish placed on a single finger on their dominant hand (gel on one finger and regular polish on another). A third finger will be left bare to serve as a control. On day 1-3 after nail polish application, the participant will have cotton swab samples taken from underneath their nail and over their nail bed, on each of the two polished nails, as well as the adjacent bare nail. These bacterial samples will be collected both before and after scrubbing (utilizing a nail pick, scrub brush, and chlorhexidine). This process will be repeat on day 5-7 after nail polish application. These samples will then be assessed for bacterial colonies in the Microbiology laboratory. Participant variables will be recorded in RedCap (scrubbing frequency, % of chipping in nails (in quartiles: 0, < 25%, < 50%, <75%, >75%, Gender, Age, Level of training, Specialty, Type of polish, Dominant hand, Duration since application of polish, Nail length in mm, Race, BMI, Type of bacteria isolated from samples).

Summary of Study Visits:

Day 0 Participants will have polish applied on two fingers on their dominant hand, one with gel polish and one with regular polish.

Day 1-3 The participants will return for their first swabs. Bacterial swabs will be obtained from the nail bed and under the fingernail of 3 fingers: the regular polish nail, the gel polish nail and a bare nail adjacent to the two polished nails, before and after a standard 5-minute scrub with chlorhexidine.

Day 5-7 The participants will return for the same procedure described above. The nail polish can be removed after this intervention. No further follow-up or involvement for participants

ELIGIBILITY:
Inclusion Criteria:

* Healthcare provider who provides patient care

Exclusion Criteria:

* Active dermatitis or other skin abnormality
* Allergy to chlorhexidine scrub soap

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Bacterial Counts Before Scrubbing Day 1-3 | 1-3 days after polish application
  Bacterial colony counts will be measured from each swab obtained from the three types of fingernails (regular polish, gel polish, bare nail).
Bacterial Counts After Scrubbing Day 1-3 | 1-3 days after polish application
  Bacterial colony counts will be measured from each swab obtained from the three types of fingernails (regular polish, gel polish, bare nail).
Bacterial Counts Before Scrubbing Day 5-7 | 5-7 days after polish application
  Bacterial colony counts will be measured from each swab obtained from the three types of fingernails (regular polish, gel polish, bare nail).
Bacterial Counts After Scrubbing Day 5-7 | 5-7 days after polish application
  Bacterial colony counts will be measured from each swab obtained from the three types of fingernails (regular polish, gel polish, bare nail).

SECONDARY OUTCOMES:
Percent of nail polish flaking (%) Day 1-3 | 1-3 days after polish application
  Percent of nail polish flaking (%) will be measured for each type of polish
Percent of nail polish flaking (%) Day 5-7 | 5-7 days after polish application
  Percent of nail polish flaking (%) will be measured for each type of polish
Nail growth (mm) Day 1-3 | 1-3 days after polish application
  Nail growth (mm) will be measured for each group
Nail growth (mm) Day 5-7 | 5-7 days after polish application
  Nail growth (mm) will be measured for each group

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Geller, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication, provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
  PI may request authorship on shared data.
Time Frame: The data will be available beginning 12 mos following publication and ending 24 months after publication.
Access Criteria: Following approval from an appropriate review board as described above and execution of a data use/sharing agreement with UNC-Chapel Hill